CLINICAL TRIAL: NCT06265948
Title: Comparsion Between Intravenous Infusion of Ketofol and Inhalational Anasthetics in Abdominal Cancer Surgeries for Post Operative Analgesia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Hussein Khalefa, doctor, Assiut University
Other Study IDs: comparsion drugs in cancer
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Abdominal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The sample will be randomly assigned into one of two equal groups ((Group-I (n: Sample size calculation was carried out using G*Power 3 software (Faul et al., 2007)1 calculated minimum sample of 80 patient candidate for cancer surgery will be needed.
  The sample will be randomly assigned into one of two equal groups ((Group-I (n=40):
  will receive standard general anesthesia as control, and Group III (n=40): will receive
  Ketofol in addition to the standard general anesthesia. The calculated sample will be
  needed to detect an effect size of 0.1
  in the RM-ANOVA (within group-between groups
  and interaction) on repeated measurements (every 2-hours postoperatively) for the
  mean VAS score, with an error probability of 0.05 and 95% power.

SUMMARY:
( post operative pain between intravenous infusion ketofol and standard inhalational general anesthesia in abdominal cancer surgeries )

DETAILED DESCRIPTION:
ketofol, which is a combination of ketamine and propofol, has been increasingly used because the advantages and disadvantages of propofol and ketamine complement each other and increase their effectiveness. Recently, the use of a combination of ketamine and propofol (ketofol) as a sedative has been attracting attention in various clinical fields. Theoretically, the combination of ketamine and propofol can reduce the dose of each drug and compensate for the disadvantages of the other through the antagonistic characteristics of both drugs, resulting in beneficial results for successful sedation

. Most of the time propofol and ketamine have been used as an induction agent in adult surgical patients but propofol may cause cardiorespiratory depression while ketamine increases heart rate and arterial blood pressure. On the other hand, the clinical effects of propofol and ketamine seem to be complementary. Ketofol is most commonly used for procedural sedation hence exploring its effectiveness for induction will be paramount for the clinical care of surgical patients Inhalation anesthetics (nitrous oxide, halothane, isoflurane, desflurane, sevoflurane, most commonly used agents in practice today) are used for induction and maintenance of general anesthesia in the operating room. The volatile anesthetics (halothane, isoflurane, desflurane, and sevoflurane) are liquids at room temperature and require the use of vaporizers for inhalational administration. Nitrous Oxide is already under normal conditions of temperature and pressure. All inhalational anesthetics provide amnesia and immobility, except for nitrous oxide, which also provides analgesia. Inhaled anesthetics are commonly used in combination with IV anesthetic agents. These agents have FDA approval for use as a general anesthetic and sedation agent in the operating room. Inhaled anesthetic agents have also had use in the intensive care unit, but this is not an FDA-approved indication. The primary applications of inhaled anesthetic agents in the ICU are sedation, refractory bronchospasm, and control of status epilepticus unresponsive to anticonvulsant medications.

ELIGIBILITY:
Inclusion Criteria:

* a. Inclusion criteria:

  1. Age group 18 - 60 years old.
  2. Both gender
  3. ASA 1and 2

Exclusion Criteria:

* a. Inclusion criteria:

  1. Age group 18 - 60 years old.
  2. Both gender
  3. ASA 1and 2 b. Exclusion criteria:

  <!-- -->

  1. Patient refusal,
  2. History of cardiac or respiratory disease, psychological disorders,
  3. High risk of regurgitation or aspiration based on a history of diabetes,

     hiatus hernia, gastroesophageal reflux, and obesity,
  4. neck pathology,
  5. Predicted difficult airway (history of difficult airway, mouth opening

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion Criteria:
  * a. Inclusion criteria:
    1. Age group 18 - 60 years old.
    2. Both gender
    3. ASA 1and 2
  Exclusion Criteria:
  * a. Inclusion criteria:
    1. Age group 18 - 60 years old.
    2. Both gender
    3. ASA 1and 2 b. Exclusion criteria:
    <!-- -->
    1. Patient refusal,
    2. History of cardiac or respiratory disease, psychological disorders,
    3. High risk of regurgitation or aspiration based on a history of diabetes,
       hiatus hernia, gastroesophageal reflux, and obesity,
    4. neck pathology,
    5. Predicted difficult airway (history of difficult airway, mouth opening
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
post operative pain | two hours
  pain according to VAS score